CLINICAL TRIAL: NCT03441555
Title: Phase 1b Study of Venetoclax and Alvocidib in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Study of Venetoclax and Alvocidib in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-186; 2017-002531-42 (EudraCT Number)
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Cancer; Acute Myeloid Leukemia (AML); relapsed Acute Myeloid Leukemia; refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — venetoclax; alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax + Alvocidib (Experimental): Venetoclax administered orally once daily (QD) and Alvocidib administered as an intravenous infusion on Days 1, 2, and 3 for all 28-day treatment cycles. Different combinations of dose levels for venetoclax and alvocidib may be explored.
  Interventions: Drug: Venetoclax; Drug: Alvocidib

INTERVENTIONS:
Drug: Venetoclax — tablet, oral
  Other Names: ABT-199
Drug: Alvocidib — Intravenous
  Other Names: Flavopiridol

SUMMARY:
An open-label, dose-escalation study to assess the safety and pharmacokinetics (PK), to determine the dose limiting toxicity (DLT) and the recommended Phase 2 dose (RPTD), and to assess the preliminary efficacy of alvocidib with venetoclax when co-administered in participants with relapsed or refractory (R/R) acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Must have adequate coagulation, hematology, kidney, and liver function, per protocol.
* Diagnosis of relapsed or refractory (R/R) acute myeloid leukemia (AML)
* Meet the following disease activity criteria:
* an established, confirmed diagnosis of AML by World Health Organization criteria excluding acute promyelocytic leukemia (APL)-M3; and
* an Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* If male participant is sexually active, he must agree from day 1 through 6 months after the last dose of alvocidib or 90 days after the last dose of venetoclax, whichever is longer, to practice the protocol-specified protection.

Exclusion Criteria:

* History of any malignancy within the last 6 months except for those specified in this protocol and low-grade malignancies not requiring active treatment such as non-melanoma skin cancer, cervical intraepithelial neoplasia, or prostate cancer in situ.
* Prior allogeneic stem cell transplant within 6 months of study drug administration and no requirement for graft versus host therapy.
* History of previous enrollment in Studies NCT02993523 or NCT03069352.
* History of exposure to alvocidib or any other cyclin-dependent kinase 9 (CDK9) inhibitor.
* History of Tumor Lysis Syndrome (TLS) due to previous exposure to venetoclax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Tmax of venetoclax | Approximately 32 days after first dose of study drug
  Time to maximum plasma concentration (Tmax) of venetoclax
Clearance of Alvocidib | Approximately 32 days after first dose of study drug
  Clearance (CL) of alvocidib
AUC0-∞ of Alvocidib | Approximately 32 days after first dose of study drug
  Area under the plasma concentration-time curve from 0 to infinity (AUC0-∞) post-dose of alvocidib
Cmax of Venetoclax | Approximately 32 days after first dose of study drug
  Maximum plasma concentration (Cmax) of venetoclax
Half-life (t1/2) of Alvocidib | Approximately 32 days after first dose of study drug
  Half-life (t1/2) of alvocidib
AUC0-24 Post-dose of Venetoclax | Approximately 32 days after first dose of study drug
  Area under the plasma concentration-time curve from 0 to 24 hours (AUC24) post-dose of venetoclax.
Cmax of Alvocidib | Approximately 32 days after first dose of study drug
  Maximum plasma concentration (Cmax) of alvocidib.
AUCt Post-dose of Alvocidib | Approximately 32 days after first dose of study drug
  Area under the plasma concentration-time curve from time zero to time t (AUCt) post-dose alvocidib.
Dose Escalation Phase: Recommended Phase 2 dose (RPTD) for Venetoclax and Alvocidib | Minimum first cycle of dosing (up to 28 days)
  RPTD will be determined using available safety and pharmacokinetics data upon completion of the dose escalation phase.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | Up to approximately 8 months
  CR is defined as the proportion of participants with documented complete response (CR) based on International Working Group (IWG) criteria.
Combined CR Rate | Up to approximately 8 months
  Combined CR rate is defined as CR + CRi (CR with incomplete blood count recovery) based on IWG criteria.
Objective Response Rate (ORR) | Up to approximately 18 months
  ORR is defined as the proportion of participants with documented partial response (PR) or better based on IWG criteria.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (14):
- United States (9):
  - USC Norris Cancer Center /ID# 170844, Los Angeles, California
  - UC Irvine /ID# 201093, Orange, California
  - University of California, Davis Comprehensive Cancer Center /ID# 170799, Sacramento, California
  - Sylvester Comprehensive Cancer /ID# 170761, Miami, Florida
  - Indiana Blood & Marrow Transpl /ID# 170793, Indianapolis, Indiana
  - NYU Langone Medical Center /ID# 201559, New York, New York
  - Weill Cornell Medical College /ID# 170800, New York, New York
  - Duke University Medical Center /ID# 170842, Durham, North Carolina
  - University of Pittsburgh Medic /ID# 170790, Pittsburgh, Pennsylvania
- Germany (2):
  - Universitaetsklinikum Dresden /ID# 168636, Dresden
  - Univ Klinik Eppendorf Hamburg /ID# 168633, Hamburg
- United Kingdom (3):
  - University Hospital of Wales /ID# 202302, Cardiff
  - Ninewells Hospital /ID# 202304, Dundee
  - St. James University Hospital /ID# 202303, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/search-results/?SearchTerm=NCT03441555&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&GenderDescriptions=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&hasResults=&isHighValue=&SortField=&SortOrder=